CLINICAL TRIAL: NCT02848105
Title: Phase II Study of Valproic Acid With Methylprenisonlone for the Treatment of Grade II-IV Acute GVHD in Patients After Allogeneic Stem Cell Transplantation
Brief Title: Valproic Acid With Methylprenisonlone for the Treatment of Acute GVHD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiong HU, Head, Blood and Marrow Transplantation Program, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJH-aGVHD-2016
Record Dates: First submitted 2016-07-26; First posted 2016-07-28 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Peripheral Blood Stem Cell Transplantation; aGVHD
Keywords: aGVHD; valproic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VPA+Methyl (Experimental): VPA added to standard methylpredisonlone treatment for aGVHD
  Interventions: Drug: VPA

INTERVENTIONS:
Drug: VPA — Valproic acid with 1000mg loading dose with 500mg q12 4 hours later to maintain a trough level above 75ug/ml

SUMMARY:
aGVHD remains as complication in patients after allogeneic stem cell transplantation. Methylprednisolone at 1~2mg/kg is considered as standard first-line treatment. In recent lab study, we demonstrated that valproic acid (VPA) as histone deacetylase inhibitor can inhibit CD4+ Th1 and Th17 cells and control the aGVDH in mice model while preserve the GVL effects. In this study, we tested the hypothesis that adding VPA to standard dose steroid treatment may improve the outcome of aGVHD.

DETAILED DESCRIPTION:
To evaluate the complete response rate of VPA+Methylpednisolone in patients with Grade II-IV aGVHD after allogenetic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Grade II-IV aGVHD
* No previous history of allergy to valproic acid
* No active and severe infection

Exclusion Criteria:

* Inclusion in other clinical trial
* GVHD Prophylaxis with valproic acid
* severe organ dysfunction: heart, lung, liver and kidney

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
complete response | 28 days after the treatment

SECONDARY OUTCOMES:
Overall response (complete + partial response) | 28 days after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jiong HU, M.D.,, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Blood & Marrow Transplantation Center, RuiJin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided